CLINICAL TRIAL: NCT05560230
Title: Intraoperative Clonidine for Postoperative Pain Management in Patients Undergoing Surgical Treatment for Endometriosis: a Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Intraoperative Clonidine for Postoperative Pain Management in Patients Undergoing Surgical Treatment for Endometriosis
Acronym: CLONIPAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022064017
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis; Postoperative Pain; Pain, Acute; Pain, Acute Postoperative
MeSH Terms: conditions — Endometriosis; Pain, Postoperative; Acute Pain | interventions — Clonidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 120 patients undergoing surgical treatment for endometriosis will be included in this prospective, randomized, double-blind, controlled trial with two arms: Intervention arm (clonidine 150 microgram). Control arm (isotonic saline).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and study medication will be handled by the hospital pharmacy. All research team members, caregiving clinicians and enrolled patients will be blinded to the study allocation arms and the randomisation list will be concealed until all statistical analyses are made.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidine (Experimental): A 100 ml isotonic saline will be mixed with 1 ml clonidine (150 μg). The blinded 100 ml bag including isotonic saline and clonidine 150 μg will be infused over 5-10 min., immediately after intubation.
  Interventions: Drug: Clonidine
- Isotonic saline (Placebo Comparator): A 100 ml isotonic saline will be mixed with 1 ml isotonic saline. The blinded 100 ml bag including isotonic saline will be infused over 5-10 min., immediately after intubation.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Clonidine — A single dose of intraoperatively administered intravenous clonidine 150 μg will be infused over 5-10 min., immediately after intubation
  Arms: Clonidine
Drug: Isotonic saline — A single dose of administered intravenous isotonic saline will be infused over 5-10 min., immediately after intubation
  Arms: Isotonic saline

SUMMARY:
The role of a single dose of intraoperative clonidine on postoperative opioid requirements, pain intensity and opioid-related side effects in patients undergoing surgical treatment for endometriosis remains scarcely explored. A prospective double-blind, randomised controlled trial investigating the effect of a single-dose of intraoperative clonidine in patients undergoing surgical treatment for endometriosis is therefore conducted.

DETAILED DESCRIPTION:
Background with aim: Acute postoperative pain is a major and common concern for the large number of patients who undergo surgery each year. Despite advances in pain management strategies, many patients continue to suffer from moderate-to-severe pain during the early postoperative period. This is concerning as unrelieved pain can result in decreased patient satisfaction, increased morbidity, prolonged hospital length-of-stay and increased risk of persistent pain. Effective treatment of acute postoperative pain should therefore be prioritized. Opioid analgesics remain the mainstay treatment for postoperative pain. The potential benefits of opioid therapy for acute pain are short-term pain control. However, there are several potential harms associated with opioid use which may outweigh the benefits including sedation, nausea, vomiting, constipation and risk of long-term use. In this respect, a single dose of clonidine could provide stable analgesia and potentially reduce the need for shorter-acting opioids. Therefore, the investigators decided to carry out the present study with the aim to examine the analgesic efficacy and safety of intraoperatively administered intravenous clonidine in patients undergoing surgical treatment for endometriosis on postoperative opioid consumption, pain intensity and opioid-related side effects.

Method: 120 patients undergoing surgical treatment for endometriosis will be included in this prospective, randomized, double-blind, controlled trial with two arms: an intervention arm (clonidine 150 microgram) and a control arm (isotonic saline). The study will be GCP-monitored, and is approved by the Danish Medicines Agency (2022064017) and the National Committee on Health Research Ethics (2209269).

Hypothesis: The investigators hypothesize that a single dose of intraoperatively administered intravenous clonidine will be effective in reducing postoperative opioid requirements, pain intensity and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

• Patients scheduled for surgical laparoscopic treatment of endometriosis at Aarhus University Hospital

Exclusion Criteria:

* Age < 18 years
* American Society of Anesthesiologists (ASA) physical status IV or V
* Allergy to clonidine
* Inability to provide informed consent
* Known severe renal insufficiency
* Known severe bradyarrhythmia
* Pregnancy, lactation:
* Daily opioid consumption the last 7 days before surgery
* Pain intensity >5 on more than half of the days during the last month

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption 0-3 hours | 3 hours after arrival at the PACU
  Opioid consumption within the first 3 hours after arrival at the PACU

SECONDARY OUTCOMES:
Cumulative opioid consumption 0-6 hours | 6 hours after arrival at the PACU
  Opioid consumption within the first 6 hours after arrival at the PACU
Pain intensity at rest | 0, 30, 60, 90 and 120 minutes after arrival at the PACU
  Pain intensity at rest (NRS; 0-10) at 0, 30, 60, 90 and 120 minutes after arrival at the PACU
Pain intensity during coughing | 0, 30, 60, 90 and 120 minutes after arrival at the PACU
  Pain intensity during coughing at 0, 30, 60, 90 and 120 minutes after arrival at the PACU
Shivering | 0, 60 and 120 minutes after arrival at the PACU
  Shivering at 0, 60 and 120 minutes after arrival at the PACU
Sedation (Ramsey Sedation Score 1-6) | 0, 60 and 120 minutes after arrival at the PACU
  Sedation at 0, 60 and 120 minutes after arrival at the PACU
PONV | 0, 60 and 120 minutes after arrival at the PACU
  Nausea and/or vomiting at 0, 60 and 120 minutes after arrival at the PACU
Discharge from the PACU | 24 hours
  Time for discharge from the PACU (hours and minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, MD, DMSc, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
The data will be shared upon reasonable request by other researchers